CLINICAL TRIAL: NCT04269720
Title: Impact of a Biofeedback Intervention on Microbiome, Metabolome, and Clinical Outcomes in Pediatric IBD
Brief Title: Biofeedback in Pediatric Inflammatory Bowel Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Ross Maltz (Other)
Responsible Party: Sponsor-Investigator, Ross Maltz, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-01100
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: IBD
Keywords: biofeedback; pediatric
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will not receive biofeedback intervention.
- Biofeedback (Experimental): Participants will receive a biofeedback intervention daily for 8 weeks. Each biofeedback session lasts approximately 10 minutes.
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback — They will also be taught how to use the biofeedback app and Inner Balance device. Additionally, they will also be educated on the principles of biofeedback and its benefits and taught how to maximize HRV by using self-regulation breathing techniques, guided imagery, and/ or self-talk.They will be given an Inner Balance device, which is an ear sensor that connects to an apple device that measures heart rate variability (HRV) and gives them access to an app that is designed to help them improve their HRV. They will be asked to use this device daily for 10 mins for the duration of the 8-week intervention. Patients and the research coordinator will have access to all of their sessions and results. The research coordinator will monitor compliance via the Heartcloud associated with their device and encourage adherence throughout the 8-week biofeedback intervention.
  Other Names: Inner Balance
  Arms: Biofeedback

SUMMARY:
This prospective, randomized, longitudinal, controlled project will occur in two phases. Phase 1 is the pre-diagnosis data collection for treatment-naïve participants who are referred for a diagnostic endoscopy/colonoscopy due to suspicion of IBD. Phase 2 (RCT) is only for patients who are diagnosed with IBD. These patients will be randomized to receive biofeedback intervention daily for 8 weeks or no biofeedback intervention. All participants will receive physician directed standard of care treatment.

DETAILED DESCRIPTION:
The inflammatory bowel diseases (IBD), which include Crohn's disease (CD) and ulcerative colitis (UC), affects 3 million Americans. In approximately 25-30% of patients, onset of these chronic diseases occurs prior to the age of 20. Despite medical advances in new therapies, the clinical remission rate on biologics is less than 50% and a significant number of patients will lose response to anti-TNF therapy over time. In addition, patients that require a change in therapy will have a lower response rate to a different biologic. Additional therapies and mechanisms that affect disease activity need to be investigated to identify complimentary treatments that can further impact remission rates without increasing side effects such as lymphoma.

Environmental factors, such as stressor exposure, can exacerbate mucosal inflammation. Patients with IBD report a lower quality of life, as well as increased anxiety and depression. Psychological interventions may improve disease activity. This study will test, using a randomized clinical trial (RCT) design, whether biofeedback intervention will attenuate disease activity. If efficacious, this study will provide a rationale for establishing biofeedback as a complimentary therapy to standard of care to ameliorate stress-induced increases in chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for Phase 1 are:

1. Age 8-17 years
2. Referred for a diagnostic colonoscopy with strong clinical concern for IBD
3. Live within a 2 hour drive of NCH

There is one additional inclusion criterion for Phase 2:

1. Patients have been diagnosed with IBD

Exclusion Criteria:

1. Participants are excluded if they have a comorbid chronic illness, perianal disease, current corticosteroid treatment, taking antibiotics within the last 3 months, psychological disorders that they are undergoing treatment or taking medication for at that time, or undergoing psychological treatments such as cognitive behavioral therapy, mindfulness, or biofeedback therapy at the time of enrollment.
2. Age and language are limited by the demands of the study (questionnaire completion)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Crohn's disease mucosal healing | pre-diagnosis to 12 month follow up
  Simple endoscopic score for CD (SES-CD) scores ileum, right colon, transverse, left colon, and rectum for the degree of ulceration. Scale ranges from 0-3, total score is calculated from sum of all variables for all 5 locations. Scores range from 0-60. Higher scores indicate worse inflammation.
Ulcerative Colitis Mucosal healing | pre-diagnosis to 12 month follow up
  Mayo endoscopic scores for the degree of ulceration. Scores range from 0-3. Higher scores indicate worse inflammation.
Disease activity( Fecal calprotectin) | pre diagnosis to 12 month follow up
  Fecal calprotectin levels from stool
Disease Activity (Crohn's disease) | pre diagnosis to 12 month follow up
  Pediatric Crohn's Disease Activity Index total score. A standard measure of disease severity that is comprised of information obtained from patient recall (pain severity, stool frequency, limitation of activities), examination (weight, height, abdominal tenderness, perirectal disease, extra- intestinal manifestations), and laboratory data. The Pediatric Crohn's Disease Activity Index total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up. Higher scores indicate more severe disease. Scores range from 0-100.
Disease Activity ( Ulcerative Colitis) | pre diagnosis to 12 month follow up
  Pediatric Ulcerative Colitis Activity Index total score. A standard Pediatric Ulcerative Colitis Activity Index. a standard measure of disease severity that is comprised pain severity, stool frequency and consistency, rectal bleeding, nocturnal bowel movements, and limitation of activities. The Pediatric Ulcerative Colitis Activity Index total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up. Higher scores indicate more severe disease. Scores range from 0-85.
Stress | pre-diagnosis to 12 month follow up
  PROMIS Pediatric Psychological Stress Experiences.Scores range from 0-60, with higher scores indicating higher levels of stress.Total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up.
Anxiety | pre-diagnosis to 12 month follow up
  PROMIS Pediatric Anxiety Short Form. Scores range from 0-60, with higher scores indicating higher levels of anxiety. Total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up.
Pediatric Quality of life | pre-diagnosis to 12 month follow up
  PedsQL. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up.
Depression | pre-diagnosis to 12 month follow up.
  Children's Depression Inventory short form. Scores range from 0-54, with higher scores indicating higher levels of depression. Total score will be used from pre-diagnosis, post-intervention, 4 months post-intervention, and 12 month follow up.

SECONDARY OUTCOMES:
Stress-related changes in the microbiome | pre diagnosis to 12 month follow up
  Microbiome α and β-diversity will be examined at pre-diagnosis, post-intervention, 4 month post-intervention, and 12 month follow-up to determine possible relationships between overall community structure between participants that received the intervention of biofeedback vs participants that were controls.
Stress-related changes in the metabolome. | pre diagnosis to 12 month follow up
  Random Forest (RF) and Boruta feature selection will be used from pre-diagnosis, post-intervention, 4 month post-intervention, and 12 month follow-up to identify metabolites and microbes.To further interpret the biological function of predictive metabolites, pathway enrichment analysis will be performed using the RaMP database, which integrates biological pathway and metabolite annotions from multiple sources (e.g. HMDB, KEGG, REACTOME, WikiPathways).

CONTACTS AND LOCATIONS:
Overall Officials: Ross Maltz, MD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No